CLINICAL TRIAL: NCT01135355
Title: Cytokine Assay for Early Identification of Pediatric Stem Cell Transplant Recipients at Risk for Respiratory Failure
Brief Title: Cytokine Assay for Early Identification of Pediatric Stem Cell Transplant Recipients
Status: Terminated | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Rajni Agarwal, Associate Professor of Pediatrics, Stanford University
Other Study IDs: PEDSBMT199; SU-09222008-1301 (Other: Stanford University); PEDSHSCT0002 (Other: Stanford University - Previous OnCore ID); 14862 (Other: stanford IRB)
Record Dates: First submitted 2010-06-01; First posted 2010-06-02 (Estimated); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Blood Stem Cell Transplant Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of our study is to determine whether a clinically relevant laboratory measurement (of seven specific immunologic biochemicals in the blood) can identify which bone marrow transplant recipients are likely to progress to respiratory failure. Our ultimate goal is to devise a comprehensive and inclusive laboratory test that is effective at determining who is likely to go on to respiratory failure, in order to facilitate early medical intervention.

ELIGIBILITY:
Inclusion Criteria:- Hematopoietic stem cell transplantation (HSCT) for any indication.

* Patients will range from age 0 to age 21. There is no gender restriction. We expect the male to female ratio to end up being about 50/50
* Ability to understand and the willingness to sign a written informed consent document.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Hematopoietic stem cell transplantation (HSCT) for any indication.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2008-07; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Compute median flourescence intensity, standard curves, and estimated pg/mL for each cytokine. | weekly during hospitalization for transplant

CONTACTS AND LOCATIONS:
Overall Officials: Rajni Agarwal-Hashmi, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States